CLINICAL TRIAL: NCT05305625
Title: Effect of Remote Ischemic Postcondioning on Glymphatic System in Acute Ischemic Stroke
Brief Title: Effect of Remote Ischemic Postcondioning on Glymphatic System in Acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XYFY2022-KL026
Record Dates: First submitted 2022-01-25; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard therapy (Experimental): Patients will be treated with Guideline standard
  Interventions: Drug: standard therapy
- remote ischemic postcondioning and standard therapy (Experimental): Patients will be treated with remote ischemic postcondioning and Guideline standard , remote ischemic postcondioning twice a day for a total of 3 days.
  Interventions: Procedure: remote ischemic postcondioning; Drug: standard therapy

INTERVENTIONS:
Procedure: remote ischemic postcondioning — remote ischemic postcondioning twice daily, for three consecutive days，the upper arm of the lighter paralyzed side was pressurized to 200mmHg, pressurized 5min and relaxed for 5 minutes for 4 cycles as a complete remote ischemic postcondioning
  Arms: remote ischemic postcondioning and standard therapy
Drug: standard therapy — received standardized treatment

SUMMARY:
Investigators aimed to investigate the changes of glymphatic function after remote ischemic postcondioning treatment in acute ischemic stroke .

ELIGIBILITY:
Inclusion Criteria:

* The patient was 18-80 years old;
* The NIHSS score was ≤ 25 and NIHSS > 5，Glasgow coma score ≥ 8;
* The patients were diagnosed as anterior circulation cerebral infarction and could start remote ischemic postcondioning within 24 hours after onset
* Normal to random time within 24 hours
* Written informed consent signed by patients or their families

Exclusion criteria:

* patients receiving thrombolysis or endovascular therapy;
* modified Rankin scale (mRS) score ≥ 2 before this attack;
* other intracranial lesions, such as cerebral hemorrhage, cerebral venous disease, severe subclavian artery stenosis and other diseases involving the brain;
* Arterial blood pressure ≤ 90/60mmHg or ≥ 180/100mmHg after treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes of glial lymphatic system | from baseline to 3 day
  The size of the vascular spaces was assessed by brain magnetic resonance of ischemic postcondioning group and standard therapy group

SECONDARY OUTCOMES:
Differential expression pattern of differential proteins | from baseline to 3 day
  Differential expression pattern of differential proteins in blood of patients with remote ischemic postcondioning group and standard therapy group

IPD SHARING:
Plan to Share IPD: No